CLINICAL TRIAL: NCT01550380
Title: A Study of BKM120 as a Single Agent in First Line Therapy in Advanced, Metastatic, or Recurrent Endometrial Cancers
Brief Title: BKM120 in Advanced, Metastatic, or Recurrent Endometrial Cancers
Acronym: BKM120
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI47841
Record Dates: First submitted 2011-07-13; First posted 2012-03-12 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — NVP-BKM120 (BKM120) is an oral pan-class I phosphatidylinositol-3-kinase (PI3K) inhibitor belonging to the 2,6-dimorpholino pyrimidine derivative family.Supplied in 10mg or 50mg capsules. Starting dose: 100mg Once Daily
  Other Names: 5-[2,6-Di(4-morpholinyl)-4-pyrimidinyl]-4-(trifluoromethyl)-2-pyridinamine

SUMMARY:
This is a phase II open label fixed dose study in subjects with advanced, metastatic, or refractory endometrial or ovarian, fallopian tube, or primary peritoneal cancer with PI3 kinase pathway activation as demonstrated by PIK3CA gene mutation, PTEN gene mutation, or PTEN null/low protein expression.

DETAILED DESCRIPTION:
Given the mechanisms of action and the safety profiles and tolerability of BKM120 (NVP-BKM120), the use of this agent may provide benefit to patients with endometrial and ovarian cancer. Endometrial and ovarian cancer are leading causes of cancer death in women and there are limited treatment options for those with metastatic or refractory disease. Alterations of the PI3K/PTEN/Akt pathway have been identified in many cancers, including endometrial and ovarian cancers. Tumors with PI3K mutations have demonstrated sensitivity to this compound therefore justifying use of this agent in subjects with endometrial or ovarian, fallopian tube, or primary peritoneal cancer. Therefore use of this agent in cancer patients with PI3 kinase pathway activation offers a reasonable treatment option.

Patients will be initially treated with single agent BKM120 for 28 days at a dose of 100mg per day. CT response will be adjudged post BKM120 therapy at day 28. If there is no significant progression on CT scan, patients will be continued on BKM120 for another two cycles (28 days per cycle [+/- 3 days]). Response assessments will then be done at that time (after the third 28 day cycle). If there is no significant progression on CT scan, then the patients will continue BKM120 with response assessments using standard CT criteria every two cycles (28 days per cycle [+/- 3 days]) thereafter.

If disease progression is observed, patient will have completed the study. Patient will be seen within 30 days for end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced, metastatic, recurrent, or persistent endometrial or ovarian, fallopian tube, or primary peritoneal cancer.
* Tumor must demonstrate PI3 Kinase pathway activation: defined as PIK3CA gene mutation, PTEN gene mutation, or PTEN null/low protein expression.
* Prior therapy:

  * Patients must not have had cytotoxic therapy directed at metastatic disease. Adjuvant chemotherapy is permitted.
  * Patients must NOT have received any non-cytotoxic therapy for metastatic or recurrent disease, except for hormonal therapy or immunologic therapy.
  * Patients with persistent or refractory disease after upfront surgery and adjuvant chemotherapy are eligible.
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Patients must have at least one site of measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 for solid tumors or the appropriate disease classification/criteria for the target population)
* Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
* Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium ≥ the lower limit of normal
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present)
* Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome)
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
* Serum amylase ≤ ULN
* Serum lipase ≤ ULN
* Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
* INR ≤ 2
* Able to provide informed consent & have signed an approved consent form that conforms to federal & institutional guidelines.

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor.
* Patients with a known hypersensitivity to BKM120 or to its excipients.
* Patients with untreated brain metastases are excluded. However, patients with metastatic Central Nervous System (CNS) tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (including radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy (other than stable low dose corticosteroid therapy as outlined in exclusion criteria #14).
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
  * Meets the cut-off score of ≥ 10 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9) will be excluded from the study unless overruled by the psychiatric assessment
* Patients with diarrhea ≥ CTCAE grade 2

  • If patient is treated for diarrhea and it resolves to grade 1, patient may be enrolled.
* Patient has active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc > 480 msec on screening ECG (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infraction within the last 6 months, documents by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documents congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that, in the opinion of the investigator, could cause unacceptable safety risks or compromise compliance with the protocol

  • Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug. Please refer to table 4-8 for a list of prohibited QT prolonging drugs with risk of Torsades de Pointes.
* Patients receiving chronic treatment with steroids or another immunosuppressive agent.

  • Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intr-articular) are allowed. Patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (e,g dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible.
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits.
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Table 4-0 for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed).
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug or whose side effects have not recovered to a grade 1 before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control. Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment.

  * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the treatment for 5 T1/2 (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation). The highly effective contraception is defined as either:

    1. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    2. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that patient.
    4. Use of a combination of any two of the following (a+b):

       * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
       * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
  * Fertile males, defined as all males physiologically capable of conceiving offspring must use condom during treatment, for 5 T1/2 (8 days) after stopping treatment and for additional 12 weeks (3 months in total after study drug discontinuation) and should not father a child in this period.
* Known diagnosis of human immunodeficiency virus (HIV) infection
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Response Rates of BKM120 | Up to 20 months
  1. To assess response rate in patients with endometrial cancer treated with first line BKM120.
  2. To assess response rate in patients with ovarian, fallopian tube, and primary peritoneal cancer treated with first line BKM120.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 20 months
  1. To determine the progression free survival (PFS) in patients with endometrial cancer treated with first line BKM120.
  2. To document the non-progression rate at 12 weeks in patients with endometrial cancer treated with first line BKM120.
  3. To determine the progression free survival (PFS) in patients with ovarian, fallopian tube, and primary peritoneal cancer treated with first line BKM120.
  4. To document the non-progression rate at 12 weeks in patients with ovarian, fallopian tube, and primary peritoneal cancer treated with first line BKM120.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Werner, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States